CLINICAL TRIAL: NCT02970539
Title: A Phase 1b Study of Oraxol in Combination With Ramucirumab in Patients With Gastric, Gastro-esophageal, or Esophageal Cancers
Brief Title: Ph1b Study of Oraxol in Comb. w. Ramucirumab in Patients w. Gastric, Gastro-esophageal, or Esophageal Cancers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Athenex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KX-ORAX-005
Record Dates: First submitted 2016-11-03; First posted 2016-11-22 (Estimated); Last update posted 2022-02-16 (Actual); Status verified 2021-02

CONDITIONS: Gastric Cancer; Esophageal Cancer; Gastro-esophageal Cancer
MeSH Terms: conditions — Stomach Neoplasms; Esophageal Neoplasms | interventions — Paclitaxel; Ramucirumab

STUDY DESIGN:
Intervention Model Description: Part 1 of the study will follow the standard "3+3" study design to determine the MTD of Oraxol administered continuously for 3 consecutive days per week (3-day MTD) in combination with ramucirumab. And Part 2 will obtain confirmatory activity, safety, and tolerability data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Oraxol +Ramucirumab (Experimental): Oraxol (oral HM30181 + oral paclitaxel)
  * HM30181 methanesulfonate monohydrate - supplied as 15-mg HM30181AK-US tablets
  * Paclitaxel - supplied as 30-mg capsules Ramucirumab - supplied as a solution at a concentration of 10 mg/mL
  Interventions: Drug: Oraxol; Drug: Ramucirumab

INTERVENTIONS:
Drug: Oraxol — Oraxol (Paclitaxel and HM30181A) will be dosed orally. Paclitaxel will be supplied as capsules and HM30181A will be supplied as tablets.
  Other Names: oral HM30181AK-US tablet and paclitaxel capsule
Drug: Ramucirumab — Ramucirumab will be administered by iv infusion and supplied as a solution at a concentration of 10 mg/mL
  Other Names: LY3009806

SUMMARY:
This is a nonrandomized, open-label, single group assignment, safety, tolerability and pharmacokinetic (PK) study to determine the MTD and optimal dosing regimen of Oraxol in combination with ramucirumab.

DETAILED DESCRIPTION:
This is a sequential-group, dose escalation trial to determine the maximum tolerated dose of oral Oraxol in combination with intravenous ramucirumab. After a screening period of up to 28 days subjects will be enrolled into the treatment phase of the study. Each cycle of therapy will last 4 weeks. Subjects may continue in the study until they experience disease progression or unacceptable toxicity. Three to six subjects will be enrolled at each dose level. Once the tolerability of a dose level has been determined, an additional 3-6 subjects may be enrolled at a higher dose level, to determine the maximum tolerated dose. Safety will be monitored through recording of adverse events, serious adverse events, monitoring of laboratory tests including hematology, blood chemistry, urinalyses, physical examinations and electrocardiograms. Subjects will undergo radiographic assessments for tumor response at specified time points. Blood samples will also be obtained in the first cycle of therapy at multiple time points for determination of the amount of paclitaxel and metabolites and HM30181 in the circulation. After the treatment period, there will be a follow-up period during which the subject or family may be contacted every three months for follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following criteria to be included in this study:

  1. Signed written informed consent 2. ≥18 years of age 3. Histologically or cytologically confirmed diagnosis of advanced stage gastric, gastro-esophageal (Part 1 or Part 2), or esophageal adenocarcinoma (Part 1 only) with disease progression on or after prior fluoropyrimidine- or platinum-containing chemotherapy 4. Have documented testing for HER2-neu overexpression, and for those with tumors overexpressing HER2-neu, have documented progression on Trastuzumab-containing therapy 5. Measurable disease on computed tomography (CT) scan of thorax, abdomen, and pelvis, per RECIST v1.1 criteria 6. Able to swallow oral medication as an intact dosage form 7. Adequate hematologic status as demonstrated by not requiring transfusion support or granulocyte-colony stimulating factor (G-CSF) to maintain:
  * ANC ≥1500 cells/mm3
  * Platelet count ≥100 x 109/L
  * Hemoglobin ≥10 g/dL; subjects with thalassemia having a hemoglobin <10 g/dL may be enrolled, per Investigator discretion 8. Adequate liver function as demonstrated by:
  * Total bilirubin of ≤1.5 mg/dL
  * Alanine aminotransferase (ALT) ≤3 x upper limit of normal (ULN) or ≤5 x ULN if liver metastasis is present
  * Alkaline phosphatase ≤3 x ULN or ≤5 x ULN if bone or liver metastasis is present
  * Gamma-glutamyl transferase (GGT) <10 x ULN 9. Adequate renal function as demonstrated by:
  * Serum creatinine ≤1.5 x ULN or creatinine clearance calculation ≥60 mL/min as calculated by the Cockcroft and Gault formula
  * Urinary protein ≤1+. If urinary protein is ≥2+, a 24-hour urine collection for protein must demonstrate <1000 mg of protein in 24 hours to allow participation in this protocol.

    10. Normal prothrombin time (PT) or international normalized ratio (INR) and normal activated partial thromboplastin time (aPTT) unless subject is on anticoagulation therapy 11. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 12. Life expectancy of at least 3 months 13. Women must be postmenopausal (>12 months without menses) or surgically sterile (ie, by hysterectomy and/or bilateral oophorectomy) or must be using effective contraception (ie, oral contraceptives, intrauterine device, double barrier method of condom and spermicide) and agree to continue use of contraception for 30 days after their last dose of study drug.

    14. Sexually active male subjects must use a barrier method of contraception during the study and agree to continue the use of male contraception for at least 30 days after the last dose of study drug.

Exclusion Criteria

Subjects who meet any of the following criteria will be excluded from this study:

1. Unresolved toxicity from previous anticancer treatments, including investigational products (subjects must have recovered all unacceptable toxicity to ≤ Grade 1 Common Terminology Criteria for Adverse Events [CTCAE] toxicity). This does not extend to symptoms or findings that are attributable to the underlying disease.
2. Received investigational products within 14 days or 5 half-lives of the first study dosing day, whichever is longer; subjects receiving biologic agents (eg, monoclonal antibodies) require a 30-day washout period.
3. Are currently receiving other medications or radiation intended for the treatment of their malignancy
4. Central nervous system metastases, including leptomeningeal involvement
5. Women of childbearing potential who are pregnant or breastfeeding
6. Currently taking a concomitant medication, other than a premedication, that is:

   * A strong P-glycoprotein (P-gp) inhibitor or inducer. Subjects who are taking such medications but who are otherwise eligible may be enrolled if they discontinue the medication ≥1 week before dosing
   * An oral medication with a narrow therapeutic index known to be a P-gp substrate within 24 hours prior to start of dosing in the study
   * Medications known to be strong inhibitors (gemfibrozil) or inducers (rifampin) of cytochrome P450 (CYP) 2C8 or medications known to be strong CYP3A4 inhibitors (eg, ketoconazole) or inducers (eg, rifampin or St. John's Wort). Subjects who are currently taking such medications but who are otherwise eligible may be enrolled if they discontinue the medication 1 week before dosing and remain off that medication during treatment with Oraxol.
7. Use of warfarin. Participants receiving warfarin who are otherwise eligible and who may be appropriately managed with low molecular weight heparin, in the opinion of the Investigator, may be enrolled in the study provided they are switched to low molecular weight heparin at least 7 days prior to receiving study treatment.
8. Require chronic use of nonsteroidal anti-inflammatory drugs (NSAIDs), chronic antiplatelet therapy, dipyridamole, clopidogrel, or similar agents. Aspirin up to 325 mg per day is allowed.
9. Unable to receive iv contrast for required CT scans
10. Poorly-controlled hypertension (>160 mm Hg systolic or >100 mm Hg diastolic for >4 weeks) despite standard medical management. Subjects may be rescreened after adjustment of their antihypertensive medication.
11. Serious or nonhealing wound, ulcer, or bone fracture within 28 days prior to first dose of protocol therapy
12. Prior history of GI perforation/fistula (within 6 months of first dose of protocol therapy) or risk factors for perforation
13. Grade 3 or 4 GI bleeding within 3 months prior to first dose of protocol therapy
14. Arterial thromboembolic event including, but not limited to, myocardial infarction, transient ischemic attack, cerebrovascular accident, or unstable angina within 6 months prior to first dose of protocol therapy
15. Deep vein thrombosis (DVT) or pulmonary embolus or any other significant thromboembolic event during the 3 months prior to first dose of protocol therapy
16. Child-Pugh Class B or C cirrhosis of the liver or cirrhosis (any degree) and a history of hepatic encephalopathy or a history of ascites resulting from cirrhosis requiring diuretics or paracentesis
17. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, poorly controlled diabetes or diabetes with established vascular complications, chronic pulmonary disease requiring oxygen, known bleeding disorders, or any concomitant illness or social situation that would limit compliance with study requirements
18. Medical condition that, in the opinion of the investigator, may interfere with oral drug absorption
19. Major surgery within 28 days prior to first dose of protocol therapy, or minor surgery/subcutaneous venous access device placement within 7 days prior to the first dose of protocol therapy, or elective or major surgery planned to be performed during the course of the clinical trial
20. History of hypersensitivity to paclitaxel, not attributed to a hypersensitivity type reaction to Cremophor®, or history of hypersensitivity type reaction to polysorbate 80 or other components of the formulation of Oraxol
21. History of developing any condition during prior treatment with ramucirumab for which ramucirumab must be permanently discontinued according to the ramucirumab Investigator's Brochure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-12-08 (Actual); Primary Completion 2019-03-27 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | The first 4 weeks
  The primary endpoint of determining the MTD will be based on DLT

SECONDARY OUTCOMES:
To determine the safety and tolerability of Oraxol in combination with ramucirumab | through study completion
  Safety assessments will consist of determining and recording all AEs (including for both increasing and decreasing severity) and SAEs
The recommended Phase 2 dose of Oraxol in combination with ramucirumab | One month
  Evaluation of the 3-day MTD for Oraxol in combination with ramucirumab, including safety, tolerability, and pharmacokinetics, will be used to determine the recommended Phase 2 dose
To characterize the area under the blood concentration curve (AUCt) of Oraxol in combination with ramucirumab | Day 1 and 3: Predose, 8 timepoints up to 8 hours postdose; Day 2: Predose; Day 8 and 15: Predose, and between 1 and 3 hours postdose
  Derived by noncompartmental analysis using the plasma concentration-time data of Oraxol (paclitaxel and its major metabolites, 3'-p-hydroxy paclitaxel and 6α-hydroxy paclitaxel, and HM30181 methanesulfonate monohydrate and its M1 metabolite)
To characterize the area under the plasma concentration-time curve from 0 to 8 hours (AUC0-8h) of Oraxol in combination with ramucirumab | Day 1 and 3: Predose, 8 timepoints up to 8 hours postdose; Day 2: Predose; Day 8 and 15: Predose, and between 1 and 3 hours postdose
  Derived by noncompartmental analysis using the plasma concentration-time data of Oraxol (paclitaxel and its major metabolites, 3'-p-hydroxy paclitaxel and 6α-hydroxy paclitaxel, and HM30181 methanesulfonate monohydrate and its M1 metabolite)
To characterize the maximum observed plasma concentration (Cmax) of Oraxol in combination with ramucirumab | Day 1 and 3: Predose, 8 timepoints up to 8 hours postdose; Day 2: Predose; Day 8 and 15: Predose, and between 1 and 3 hours postdose
  Derived by noncompartmental analysis using the plasma concentration-time data of Oraxol (paclitaxel and its major metabolites, 3'-p-hydroxy paclitaxel and 6α-hydroxy paclitaxel, and HM30181 methanesulfonate monohydrate and its M1 metabolite)
To characterize the minimum observed plasma concentration (Cmin) of Oraxol in combination with ramucirumab | Day 1 and 3: Predose, 8 timepoints up to 8 hours postdose; Day 2: Predose; Day 8 and 15: Predose, and between 1 and 3 hours postdose
  Derived by noncompartmental analysis using the plasma concentration-time data of Oraxol (paclitaxel and its major metabolites, 3'-p-hydroxy paclitaxel and 6α-hydroxy paclitaxel, and HM30181 methanesulfonate monohydrate and its M1 metabolite)
To characterize the plasma half-life (t1/2) of Oraxol in combination with ramucirumab | Day 1 and 3: Predose, 8 timepoints up to 8 hours postdose; Day 2: Predose; Day 8 and 15: Predose, and between 1 and 3 hours postdose
  Derived by noncompartmental analysis using the plasma concentration-time data of Oraxol (paclitaxel and its major metabolites, 3'-p-hydroxy paclitaxel and 6α-hydroxy paclitaxel, and HM30181 methanesulfonate monohydrate and its M1 metabolite)
To characterize the accumulation factor (R) of Oraxol in combination with ramucirumab | Day 1 and 3: Predose, 8 timepoints up to 8 hours postdose; Day 2: Predose; Day 8 and 15: Predose, and between 1 and 3 hours postdose
  Derived by noncompartmental analysis using the plasma concentration-time data of Oraxol (paclitaxel and its major metabolites, 3'-p-hydroxy paclitaxel and 6α-hydroxy paclitaxel, and HM30181 methanesulfonate monohydrate and its M1 metabolite)
To characterize the apparent volume of distribution (Vd/F) of Oraxol in combination with ramucirumab | Day 1 and 3: Predose, 8 timepoints up to 8 hours postdose; Day 2: Predose; Day 8 and 15: Predose, and between 1 and 3 hours postdose
  Derived by noncompartmental analysis using the plasma concentration-time data of Oraxol (paclitaxel and its major metabolites, 3'-p-hydroxy paclitaxel and 6α-hydroxy paclitaxel, and HM30181 methanesulfonate monohydrate and its M1 metabolite)
To characterize the apparent total clearance (CL/F) of Oraxol in combination with ramucirumab | Day 1 and 3: Predose, 8 timepoints up to 8 hours postdose; Day 2: Predose; Day 8 and 15: Predose, and between 1 and 3 hours postdose
  Derived by noncompartmental analysis using the plasma concentration-time data of Oraxol (paclitaxel and its major metabolites, 3'-p-hydroxy paclitaxel and 6α-hydroxy paclitaxel, and HM30181 methanesulfonate monohydrate and its M1 metabolite)
Preliminary activity of Oraxol plus ramucirumab as determined by response rate | Subjects will be evaluated for tumor response per RECIST v1.1 criteria after every 8 weeks (ie, at Weeks 9, 17, 25, etc).
  Tumor response will be evaluated according to RECIST v1.1 criteria
Preliminary activity of Oraxol plus ramucirumab as determined by progression-free survival | Subjects will be evaluated for tumor response per RECIST v1.1 criteria after every 8 weeks (ie, at Weeks 9, 17, 25, etc).
  Tumor response will be evaluated according to RECIST v1.1 criteria
Preliminary activity of Oraxol plus ramucirumab as determined by overall survival | Investigator,telephone, or family member contact or public records access will be performed every 3 months for the purpose of assessing overall survival.
  There will be a Follow-up Period during which survival data will be collected

CONTACTS AND LOCATIONS:
Overall Officials: David Cutler, MD, Study Director — Athenex, Inc.
Locations (5):
- CTRC-UT, San Antonio, Texas, United States
- Taiwan (4):
  - China Medical University Hospital, Taichung
  - Tri-Service General Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Lotung Poh-Ai Hospital, Yilan

IPD SHARING:
Plan to Share IPD: No